CLINICAL TRIAL: NCT01644227
Title: Dual Mobility Cup in Total Hip Arthroplasty Preventing Dislocation in Patients at Risk
Status: Completed | Type: Observational
Sponsor: Sundsvall Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Sebastian-1
Record Dates: First submitted 2012-06-24; First posted 2012-07-19 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2015-10

CONDITIONS: Femoral Neck Fracture; Osteoarthritis
Keywords: Hip surgery; dual mobility cup; dislocation; total hip arthroplasty
MeSH Terms: conditions — Femoral Neck Fractures; Osteoarthritis; Joint Dislocations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Retrospectively study reviewing 34 patients operated with dual mobility cups in total hip arthroplasty between January 2009 and June 2012 at Sundsvall Hospital.

Hypothesis: The dual mobility socket reduce the rate of dislocation in patient at high risk but increase the incidence of postoperative infection.

DETAILED DESCRIPTION:
Retrospectively study reviewing 34 patients operated with dual mobility cups in total hip arthroplasty between January 2009 and June 2012 at Sundsvall Hospital.

Indications for surgery is recurrent dislocation or patients at risk for dislocation after total hip arthroplasty suffering osteoarthritis or femoral neck fracture.

Patients are followed recording complications, reoperations, functional outcome (Harris hip score and EQ5D) in june 2012.

ELIGIBILITY:
Inclusion Criteria:

* operated with an cemented dual mobility socket at Sundsvall hospital

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients operated with an cemented dual mobility cups at Sundsvall hospital between 2009-2012.
  Indications for surgery are recurrent dislocation and patients at risk for dislocation mainly due to comorbidity, neuromuscular, psychiatric or cognitive disorders.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2012-06; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Prosthetic dislocation | 2012 (up to 3 years postoperatively)
  Incidence of postoperative dislocations of the prosthesis

SECONDARY OUTCOMES:
Complication | 2012 (up to 3 years postoperatively)
  Incidence of complications and reoperations
Hip function | 2012 (up to 3 years postoperatively)
  Patient reported hip function; Harris hip score
Quality of life | 2012 (up to 3 years postoperatively)
  Patient reported quality of life: EQ5D

CONTACTS AND LOCATIONS:
Overall Officials: Arkan S Sayed Noor, MD, PhD, Principal Investigator — Landstinget Västernorrland
Locations (1):
- Orthopaedic department, Sundsvall, Västernorrland County, Sweden

REFERENCES:
- [Result] Mukka SS, Mahmood SS, Sjoden GO, Sayed-Noor AS. Dual mobility cups for preventing early hip arthroplasty dislocation in patients at risk: experience in a county hospital. Orthop Rev (Pavia). 2013 Jun 11;5(2):48-51. doi: 10.4081/or.2013.e10. Print 2013 Jun 7. PMID 23888200